CLINICAL TRIAL: NCT02580448
Title: A Phase 1/2 Open-Label Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy of Seviteronel in Subjects With Advanced Breast Cancer
Brief Title: CYP17 Lyase and Androgen Receptor Inhibitor Treatment With Seviteronel Trial (INO-VT-464-006; NCT02580448)
Acronym: CLARITY-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innocrin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INO-VT-464-CL-006
Record Dates: First submitted 2015-10-07; First posted 2015-10-20 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Cancer of the Breast; Breast Cancer; Advanced Breast Cancer; Metastatic Breast Cancer; Male Breast Cancer; Triple Negative Breast Cancer; ER+ Breast Cancer
Keywords: Breast Cancer; Breast; Advanced Breast Cancer; Metastatic Breast Cancer; CYP17; Male Breast Cancer; Triple Negative Cancer; ER+ Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Triple Negative Breast Neoplasms | interventions — seviteronel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Female Triple Negative Breast Cancer Patients (Experimental): TNBC Patients - Enrollment is complete in this cohort
  Interventions: Drug: Seviteronel
- Female Estrogen Receptor (+) Breast Cancer Patients (Experimental): Female ER(+) BC Patients - Enrollment is complete in this cohort
  Interventions: Drug: Seviteronel
- Male Breast Cancer Patients (Experimental): Locally advanced or metastatic males with BC
  Interventions: Drug: Seviteronel

INTERVENTIONS:
Drug: Seviteronel — Seviteronel given daily with evening meal in 28 day cycles

SUMMARY:
The goal of this clinical study is to determine the safety, pharmacokinetics, pharmacodynamics and efficacy and activity of seviteronel, a lyase-selective inhibitor of CYP17, in patients with advanced breast cancer.

DETAILED DESCRIPTION:
This is an open-label, Phase 1/2 study of seviteronel in subjects with TNBC or ER +/HER2 normal unresectable locally advanced breast cancer. Only women will be enrolled in Phase 1 and both men and women enrolled into their respective cohorts in Phase 2. There will be a dose confirmation Phase 1 portion of the study to establish the recommended Phase 2 dose (RP2D) for women with breast cancer using a non-stratified, combined cohort of women with TNBC or ER+ BC. Cohort expansion will occur in Phase 2 at the RP2D confirmed/established in Phase 1 using separate TNBC and ER+ cohorts. The Phase 2 portion of the study is divided into three parallel cohorts:

Cohort 1: Female TNBC Subjects Cohort 2: Female ER+ Subjects Cohort 3: Male ER+ BC or TNBC Subjects

ELIGIBILITY:
Inclusion Criteria

Each subject eligible to participate in this study must meet or have all the following criteria:

1. Is 18 years of age or older.
2. Can provide written informed consent or have their legal representatives provide written informed consent
3. Have documented histological or cytological evidence of invasive cancer of the breast, defined by one of the following:

   * ER+ breast cancer, defined as positive if ≥ 1% by IHC and HER2 normal, defined as IHC 0-1+ or IHC 2+(and FISH<2), or FISH < 2.0
   * TNBC, defined as ER-/PgR- if 0 % by IHC and HER2 normal, defined as IHC 0-1+ or IHC 2+(and FISH<2), or FISH < 2.0
4. ECOG PS of 0 or 1 for Females, 0, 1, or 2 for Males.
5. Undergoing or willing to undergo gonadal suppression:

   * Female subjects with ER+/HER2 normal tumors must be post-menopausal defined by local practice. Ovarian suppression with a LHRH analogue to achieve cessation of regular menses is allowed on study
   * Male subjects must be undergoing or willing to undergo gonadal suppression whilst on study drug and continue with the LHRH analogue for the duration of the study
6. Subjects must have adequate hematopoietic function as evidenced by:

   * WBC ≥ 3,000/μl
   * ANC ≥ 1,500/μl
   * Platelet count ≥ 100,000/μl
   * HGB ≥ 9 g/dl and not transfusion dependent
7. Adequate liver function, including all the following:

   * Total serum bilirubin ≤2.0 x ULN unless the subject has documented Gilbert syndrome;
   * Aspartate and alanine aminotransferase (AST & ALT) ≤3.0 x ULN or ≤5.0 x ULN if subject has liver metastasis;
   * Alkaline phosphatase ≤3.0 x ULN or ≤5 x ULN in case of bone metastasis and/or hepatic metastasis
8. Subjects must have adequate renal function as evidenced by a serum creatinine of ≤ 2.0 mg/dl.
9. Potassium (K+) ≥3.5 mEq/L
10. Women of child-bearing potential must have a negative serum or urine pregnancy test within 72 hours of C1D1.
11. Women of child-bearing potential and male subjects with a female partner of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at Screening and continuing throughout the study period and for 3 months after final study drug administration i. Two acceptable forms of birth control include:

1. Condom (barrier method of contraception), and 2. One of the following:

1. Oral, injected or implanted hormonal contraception
2. Placement of an intrauterine device (IUD) or intrauterine system (ISU)
3. Additional barrier methods of contraception: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
4. Vasectomy or surgical castration ≥ 6 months prior to Screening. 12. Able to swallow study medication 13. Able to comply with study requirements

Exclusion Criteria

1. Received any investigational agent within 5 half-lives of the agent in question; if the half-life is not known, ≤ 28 days of C1D1.
2. Received palliative radiotherapy ≤ 2 weeks of C1D1
3. Received any other therapeutic treatment for breast cancer ≤ 2 weeks of C1D1, except for hormonal therapies.
4. Symptomatic CNS metastases.
5. History of another invasive malignancy ≤ 3 years of C1D1.
6. A QTcF interval >470 msec on the Screening ECG. If the ECG QTcF interval is >470 msec, then the mean QTcF of a triplicate ECGs can be used and if the mean is <470 msec, the subject may be enrolled.
7. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, atrial fibrillation with rapid ventricular response, torsades de pointes, second degree or third degree atrioventricular heart block without a permanent pacemaker in place).
8. Class III or IV Congestive Heart Failure (CHF) as defined by the New York Heart Association (NYHA) functional classification system within the previous 6 months
9. Initiated a bone modifying agent (e.g. denosumab) ≤ 28 days of C1D1.
10. Any medical condition that could preclude their participation in the study, pose an undue medical hazard, or which could interfere with the interpretation of the study results.
11. A history of seizure ≤ 2 years of C1D1 or those who require prophylactic anti-seizure medications.
12. A history of loss of consciousness or transient ischemic attack ≤ 12 months before C1D1.
13. Known active HIV, Hepatitis B, or Hepatitis C infections.
14. Known or suspected hypersensitivity to seviteronel, or any components of the formulation.
15. Any other condition which in the opinion of the investigator would preclude participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Estimate efficacy of seviteronel as measured by clinical benefit rate at 16 weeks (CBR16) for female subjects with TNBC. | Duration of Study
Estimate efficacy of seviteronel as measured by clinical benefit rate at 24 weeks (CBR24) for female subjects with ER+ BC. | Duration of Study
Estimate efficacy of seviteronel as measured by CBR16 for all male BC subjects. | Duration of Study

SECONDARY OUTCOMES:
Describe the pharmacokinetics of seviteronel | At least monthly over the first eight 28-day cycles
  Area under the curve concentration verses time curve and Peak Plasma Concentration
Estimate efficacy of seviteronel as measured by the overall response rate (ORR) based on RECIST 1.1 | At least monthly over the first eight 28-day cycles
Estimate efficacy of seviteronel as measured by progression-free survival (PFS) | At least monthly over the first eight 28-day cycles
Describe the safety profile of seviteronel | Duration of the study
Compare the safety profile of seviteronel with or without concurrent glucocorticoid administration | Duration of the study
Compare the CBR16 with or without concurrent glucocorticoid administration for female subjects with TNBC | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Brown, BS, Study Chair — Sponsor GmbH
Locations (36):
- United States (36):
  - Wallace Tumor Institute- University of Alabama, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - University of Colorado, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists- North, St. Petersburg, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - SCRI - HCA Midwest Division, Kansas City, Kansas
  - University of Louisville Hospital / James Brown Cancer Center, Louisville, Kentucky
  - Maryland Oncology Hematology, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Masonic Cancer Center, Minneapolis, Minnesota
  - Cancer Network/Oncology Associates PC, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Memorial Sloan Kettering, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center - Oncology Research, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Oncology Hematology Care, Inc, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Charleston Hematology and Oncology Associates, Charleston, South Carolina
  - Precision Cancer Research/Brig Center for Cancer Care and Survivorship, LLC, Knoxville, Tennessee
  - SCRI Tenessee Oncology Nashville, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - The Center for Cancer and Blood Disorders (Fort Worth), Fort Worth, Texas
  - US Oncology, Fort Worth, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Oncology Associates, Norfolk, Virginia